CLINICAL TRIAL: NCT04624360
Title: Randomised Controlled Trial Comparing the Effect of Intravenous Dexamethasone vs. Placebo on the Duration of Analgesia of Spinal Anaesthesia for Caesarean Sections at the Victoria Jubilee Hospital in Jamaica
Brief Title: The Effect of IV Dexamethasone on the Duration of Analgesia of Spinal Anaesthesia for C-Sections at a Jamaican Hospital
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Collaborators: National Health Fund of Jamaica (Unknown)
Responsible Party: Principal Investigator, Renee Nesbeth, Dr., The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VJH Dexa Study
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Drug A (Experimental): Dexamethasone 8mg intravenous administration stat dose post clamping of the umbilical cord
  Interventions: Drug: Dexamethasone
- Study Drug B (Placebo Comparator): Normal saline 2cc intravenous stat dose administered after clamping of the umbilical cord
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Intravenous of Dexamethasone 8 mg post clamping of the umbilical cord
  Other Names: Study Drug A
  Arms: Study Drug A
Other: Placebo — 2cc 0.9% Saline
  Other Names: Study Drug B
  Arms: Study Drug B

SUMMARY:
Dexamethasone is one of many adjuncts tested to prolong the duration of spinal anesthesia and its analgesic effect. The intent of this, a single-site, double-blinded, randomized controlled trial, is to determine if a single intravenous (IV) 8 mg dose of Dexamethasone given after clamping of the umbilical cord at Caesarean section will prolong the duration of analgesia provided by spinal anesthesia when compared to placebo. This has the power to determine if the findings in previous studies hold true in the population of women who undergo C-sections at the Victoria Jubilee Hospital. This method does not require expert skill and equipment, as such, it can be easily implemented, with no major adverse effects in the population described and provide an effective option for multimodal analgesia.

DETAILED DESCRIPTION:
This study is being conducted in accordance with the Good Clinical Practice guidelines as enunciated in the international Conference on Harmonization (ICP/GCP) of 2016 and the Declaration of Helsinki, 2013.

Sample Size:

The sample size calculated based on a study done by Shahraki et al who studied the efficacy of intravenous Dexamethasone in prolonging the duration of Spinal Anesthesia in elective Caesarean Section in an Indian population (36).

The following values were used for the calculation of the sample size: the required value of α was 5%, β was 10%, a clinically significant difference in Visual Analogue Scale (VAS) score at 1-hour post-surgery was considered 2 and the expected standard deviation was 2.5 (36). The equation used was:

n = (Zα/2+Zβ)2 *2*σ2 / d2,

where Zα/2 is the critical value of the normal distribution at α/2 (α is 0.05), Zβ is the critical value of the normal distribution at β of 0.10. σ2 is the population variance (2.52), and d is the difference to be detected (2). The calculated sample size is 14 patients in each group. In order allow for a potential loss of data up to 10% the target sample size required would be 16 in each group.

Assumptions:

1. The population size is limited by:

   1. patient's age,
   2. gestational age,
   3. the type of birth - only Caesarian births,
   4. use of a single hospital - VJH
   5. the duration of the research of approximately 2 to 3 months.
2. As a result of item 1, when the Finite Population model is used to determine the sample size -

S = Z2 * p(p-1) / E2

1 + (Z2 * p(p-1) / E2N)

Other parameters include:

1. 95% Confidence level
2. Margin of error 5%
3. Number of live births at VJH in 2016 estimated at 8140 live births
4. Number of Caesarian births same period = 1652
5. Percent of Caesarian births (with access to in 2 to 3 months) = 3.6 to 5%

The computed sample size ranges from 53 (2 months) to 72 (3 months) The decision was made to include 30 patients in each group totaling 60 persons for the sample size for this study.

Research assistants received training in the study protocol. Presentations were made to the registration clerks, obstetricians, midwives and other nursing staff to introduce them to the study.

Recruitment The registration clerk informs the patients of the study being carried out from admission to hospital. The ward nurse, upon admitting the patient, determine if they meet the criteria and indicates same to a member of the research team. Written informed consent is obtained by an independent research assistant, once it is confirmed that the patient meets the criteria, to avoid any perception of coercion on the night before or the morning of their procedure. The patient's autonomy is respected and quality medical care will is provided for those who participate in the study as well as those who decline.

Conceptual Definition of Variables Duration of analgesia: the time from intrathecal injection to the time of the first request for analgesia or Visual Analogue Pain Scale score > 4.

Duration of motor blockade: the time from intrathecal injection to the time when the patient is able to flex their knees with free movement of their feet in any plane.

Data Collection/ Storage The data collected for research is stored in a secured area in the Anesthetic Office at the Kingston Public Hospital with access limited to the research team only. Back-up of the data is stored off-site in a locked room in the Anesthetic Office of the University Hospital of the West Indies. Each patient is assigned a study number, and strict security measures are employed to ensure maximum protection of data and the privacy of the research subjects such as password protection and anonymity of data.

If a participant decides to withdraw from the study, the data collected prior to withdrawal may be used in data analysis and the same anonymity applies. Withdrawal from the study will not affect the participant's access to quality health care.

Source Data Verification This is done by cross-referencing the data entered on the data collection forms with the patients' dockets.

Statistical Analysis The data will be managed and analyzed using Statistical Package for the Social Sciences [SPSS] version 26.0 (2019). Uni-variate, bi-variate and multi-variate analysis of the data will be done. Uni-variate analysis will include means ± standard deviation. Bi-variate analysis will include will include independent/ paired t-tests for quantitative data; Chi square test and Mann-Whitney's U test where applicable. Multi-variate analysis will include regression and other measurements where necessary. A p value of less than 0.05 will be deemed statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Victoria Jubilee Hospital in Jamaica, scheduled for non-emergent LSCS under spinal anesthesia
* Age: 18 to 45 years
* Gestational Age: 37 weeks or more
* American Society of Anesthesiologists physical status class II
* Singleton fetus

Exclusion Criteria:

* Emergent Indication for caesarean section including, but not limited to:
* Fetal distress
* Cord prolapse
* Eclampsia
* Severe pre-eclampsia
* Placental abruption
* Placenta praevia
* Multiple Gestation
* Allergy to glucocorticoids/opioids/Diclofenac Na/ local anesthetics
* Contra-indication to Spinal Anesthesia
* Gestational Diabetes or Pre-gestational Diabetes
* Asthma
* Other uncontrolled comorbidities (such as cardiac, respiratory, renal, inflammatory, endocrine disease)
* Chronic steroid use
* history of Peptic Ulcer Disease or Glaucoma
* history of chronic pain
* Illicit drug users (including marijuana)
* Any patient who requires general anesthesia secondary to failure of spinal anesthesia will also be excluded

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females undergoing operative delivery
Enrollment: 60 (Estimated)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | first 4 hours after spinal anesthesia administered
  The duration of time from the administration of drugs intrathecally for spinal anesthesia to the first request for analgesia or first time the pain score is greater than 4

CONTACTS AND LOCATIONS:
Overall Officials: Christine Stephen, MB;BS, DM, Principal Investigator — University of the West Indies
Locations (1):
- Victoria Jubilee Hospital, Kingston, Non-US/Canada, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: January 2021 - December 2028

REFERENCES:
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Carvalho B, Cohen SE, Lipman SS, Fuller A, Mathusamy AD, Macario A. Patient preferences for anesthesia outcomes associated with cesarean delivery. Anesth Analg. 2005 Oct;101(4):1182-1187. doi: 10.1213/01.ane.0000167774.36833.99. PMID 16192541
- [Background] Jadon A, Bagai R. Effective pain relief after caesarean section; Are we on the right path or still on the crossroad. Journal of Obstetric Anaesthesia and Critical Care. 2019;9(1):3-6
- [Background] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Background] Marian Knight KB, Derek Tuffnell, Hemali Jayakody,Judy Shakespeare RK, Sara Kenyon,, Kurinczuk JJ. MBRRACE-UK: Saving Lives, Improving Mothers' Care - Lessons learned to inform maternity care from the UK and Ireland Confidential Enquiries into Maternal Deaths and Morbidity 2014-16. Oxford: University of Oxford; 2018
- [Background] Jno-Baptiste B, Scarlett MD, Harding H, Ehikmetalor K: The Effect of Dexamethasone on Post-operative Opioid Requirement in Patients who Underwent Gynecology Surgery at the University Hospital in Jamaica. Journal of Anesthesia & Clinical Research. 2014;5(11):5
- [Background] Sutton CD, Carvalho B. Optimal Pain Management After Cesarean Delivery. Anesthesiol Clin. 2017 Mar;35(1):107-124. doi: 10.1016/j.anclin.2016.09.010. Epub 2016 Dec 12. PMID 28131114
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] Shalu PS, Ghodki PS. To Study the Efficacy of Intravenous Dexamethasone in Prolonging the Duration of Spinal Anesthesia in Elective Cesarean Section. Anesth Essays Res. 2017 Apr-Jun;11(2):321-325. doi: 10.4103/0259-1162.194537. PMID 28663614
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. PMID 21704871
- [Background] Liu K, Hsu CC, Chia YY. Effect of dexamethasone on postoperative emesis and pain. Br J Anaesth. 1998 Jan;80(1):85-6. doi: 10.1093/bja/80.1.85. PMID 9505784
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Mathew R, Radha KR, Hema VR. Effect of Perineural and Intravenous Dexamethasone on Duration of Analgesia in Supraclavicular Brachial Plexus Block with Bupivacaine: A Comparative Study. Anesth Essays Res. 2019 Apr-Jun;13(2):280-283. doi: 10.4103/aer.AER_15_19. PMID 31198245
- [Background] Hong JY, Han SW, Kim WO, Kim EJ, Kil HK. Effect of dexamethasone in combination with caudal analgesia on postoperative pain control in day-case paediatric orchiopexy. Br J Anaesth. 2010 Oct;105(4):506-10. doi: 10.1093/bja/aeq187. Epub 2010 Jul 20. PMID 20659915
- [Background] Shahraki AD, Feizi A, Jabalameli M, Nouri S. The effect of intravenous Dexamethasone on post-cesarean section pain and vital signs: A double-blind randomized clinical trial. J Res Pharm Pract. 2013 Jul;2(3):99-104. doi: 10.4103/2279-042X.122370. PMID 24991614
- [Background] Heesen M, Rijs K, Hilber N, Eid K, Al-Oweidi A, Rossaint R, Klimek M. Effect of intravenous dexamethasone on postoperative pain after spinal anaesthesia - a systematic review with meta-analysis and trial sequential analysis. Anaesthesia. 2019 Aug;74(8):1047-1056. doi: 10.1111/anae.14666. Epub 2019 May 6. PMID 31058317
- [Background] Maged AM, Deeb WS, Elbaradie S, Elzayat AR, Metwally AA, Hamed M, Shaker A. Comparison of local and intra venous dexamethasone on post operative pain and recovery after caeseream section. A randomized controlled trial. Taiwan J Obstet Gynecol. 2018 Jun;57(3):346-350. doi: 10.1016/j.tjog.2018.04.004. PMID 29880162
- [Background] Ituk U, Thenuwara K. The effect of a single intraoperative dose of intravenous dexamethasone 8 mg on post-cesarean delivery analgesia: a randomized controlled trial. Int J Obstet Anesth. 2018 Aug;35:57-63. doi: 10.1016/j.ijoa.2018.03.008. Epub 2018 Mar 26. PMID 29773484
- [Background] Cardoso MM, Leite AO, Santos EA, Gozzani JL, Mathias LA. Effect of dexamethasone on prevention of postoperative nausea, vomiting and pain after caesarean section: a randomised, placebo-controlled, double-blind trial. Eur J Anaesthesiol. 2013 Mar;30(3):102-5. doi: 10.1097/EJA.0b013e328356676b. PMID 23022704
- [Background] Vyvey M. Steroids as pain relief adjuvants. Can Fam Physician. 2010 Dec;56(12):1295-7, e415. PMID 21156893
- [Background] Kalogera E, Dowdy SC. Enhanced Recovery Pathway in Gynecologic Surgery: Improving Outcomes Through Evidence-Based Medicine. Obstet Gynecol Clin North Am. 2016 Sep;43(3):551-73. doi: 10.1016/j.ogc.2016.04.006. PMID 27521884
- [Background] Ituk U, Habib AS. Enhanced recovery after cesarean delivery. F1000Res. 2018 Apr 27;7:F1000 Faculty Rev-513. doi: 10.12688/f1000research.13895.1. eCollection 2018. PMID 29770203
- [Background] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Background] Committee on Obstetric Practice. Committee Opinion No. 713: Antenatal Corticosteroid Therapy for Fetal Maturation. Obstet Gynecol. 2017 Aug;130(2):e102-e109. doi: 10.1097/AOG.0000000000002237. PMID 28742678
- [Background] Brownfoot FC, Gagliardi DI, Bain E, Middleton P, Crowther CA. Different corticosteroids and regimens for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2013 Aug 29;(8):CD006764. doi: 10.1002/14651858.CD006764.pub3. PMID 23990333
- [Background] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857